CLINICAL TRIAL: NCT06110819
Title: Individual Training Given to Pregnant Women in the Earthquake Zone in Their Living Spaces, the Effect of Pregnancy Follow-up on Prenatal Comfort, Distress, Risk Perception and Birth Anxiety.
Brief Title: Individual Training Given to Pregnant Women in the Earthquake Zone in Their Living Spaces,
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate (Other Government)
Responsible Party: Principal Investigator, Mine Gokduman Keles, DR.Midwifery, Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TurkishHKahramanmara
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Pregnant Women

STUDY DESIGN:
Intervention Model Description: In line with the Prenatal Care Management Guide of the Ministry of Health, each pregnant woman will be trained and monitored during their trimester until they give birth (4 follow-ups). Pregnancy training trimesters of all participants will be given in accordance with the health guide and follow-up will be done in their living spaces. During these trainings, they will be provided with care in line with the recommendations of the Ministry of Health.
Who Masked: Outcomes Assessor
Masking Description: Analyzes will not be made by the researcher.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workgroup (Experimental): .In line with the Prenatal Care Management Guide of the Ministry of Health, each pregnant woman will be trained and monitored during their trimester until they give birth (4 follow-ups). Pregnancy training trimesters of all participants will be given in accordance with the health guide and follow-up will be done in their living spaces. During these trainings, they will be provided with care in line with the recommendations of the Ministry of Health.
  Interventions: Other: Workgroup
- Control (Other): Pregnant women will be contacted by phone and the status of their follow-up in health institutions will be questioned. During these follow-ups, training is provided and monitoring is carried out in line with the Prenatal Care Management Guide of the Ministry of Health.
  Interventions: Other: control

INTERVENTIONS:
Other: control — Pregnant women will be contacted by phone and the status of their follow-up in health institutions will be questioned. During these follow-ups, training is provided and monitoring is carried out in line with the Prenatal Care Management Guide of the Ministry of Health.
  Arms: Control
Other: Workgroup — Experimental:
  .In line with the Prenatal Care Management Guide of the Ministry of Health, each pregnant woman will be trained and monitored during their trimester until they give birth (4 follow-ups). Pregnancy training trimesters of all participants will be given in accordance with the health guide and follow-up will be done in their living spaces. During these trainings, they will be provided with care in line with the recommendations of the Ministry of Health.
  Arms: Workgroup

SUMMARY:
This study aims to evaluate the effect of individual training and pregnancy follow-up given to pregnant women in the earthquake zone in their living spaces on prenatal comfort, distress, risk perception and birth anxiety.

In the randomized controlled experimental study, data will be obtained using the Personal Information Form, Pregnant Observations and Birth Results, Prenatal Comfort Scale, Prenatal Distress Scale, Pregnancy Risk Perception Scale, Oxford Birth Anxiety Scale.

DETAILED DESCRIPTION:
In the literature, it has been reported that the earthquake had a negative impact on pregnant women, as well as material and loss of life (Amarpoor Mesrkanlou, et al. 2023; Kyozuka, et al. 2022; Nishigori, et al. 2014; Watanabe, et al. al. 2016). In the study of İlavaten Mesrkanlou et al (2023); It has also been reported that post-earthquake causes insufficient weight gain in pregnant women, decreased hemoglobin levels, and adverse birth outcomes. (Amarpoor Mesrkanlou, et al. 2023). Again, in the research of Kyozuko et al., (2022); It has been reported that pregnancy complications such as gestational hypertension, respiratory diseases and mental disorders increased in pregnant women after the earthquake (Kyozuka, et al. 2022). In their study, Mesrkanlou et al., (2023) reported postpartum depression as 21.3% in 633 pregnant women in the regions affected by the East Japan earthquake (Nishigori, et al. 2014). Watanabe, et al. (2016) reported psychological distress among pregnant women in the Miyagi region of Japan as 4.9% in their study (Watanabe, et al. 2016). In addition, the earthquake may result in negative effects during pregnancy, such as premature birth, low birth weight and hypertensive disorders. (Hawkins, et al. 2019; Lian, et al. 2020; Palmeiro-Silva, et al. 2018). As a result of the 6.3 magnitude earthquake in Christchurch, New Zealand, premature birth was reported as 6.71% in 1057 pregnant women (Hawkins, et al. 2019). In addition, in the study that examined the relationships between earthquake exposure of pregnant women and negative birth outcomes and included 73,493 women, pregnant women exposed to the earthquake had a 2% higher rate of stillbirth and 14.14% higher preterm birth compared to pregnant women not exposed to the earthquake (Lian, et al. 2020). ).

In this context, increased levels of anxiety and depression during pregnancy may affect the comfort level of the pregnant woman (Matvienko-Sikar and Dockray 2017). In addition, prenatal stress is defined as the emotional reactions of the pregnant woman in terms of physical, psychological and social changes that occur during pregnancy, birth, parenthood and baby health (O'Hara and Wisner 2014). Again, inadequate prenatal care increases perinetal stress (Gooijers and Swinnen 2014). In a study conducted in Turkey, it was reported that perinetal stress affected preterm birth the most during pregnancy (Yuksel, et al. 2014). Pregnant women are among the most vulnerable people who may need special support in the event of an earthquake. Therefore, pregnant women should be provided with stronger support after the earthquake.

For this reason, it is important to provide and maintain the care of pregnant women face to face by health professionals after the earthquake (Yamashita, et al. 2019). In addition, the education given to pregnant women is also effective in preventing premature birth and postpartum depression (Çankaya and Şimşek 2021; Dennis and Dowswell 2013). In addition, it has been reported in the literature that the satisfaction of pregnant women is increased with the different education models (home visits, medical care, individualized care) provided during pregnancy. (MOUNTAINS, et al. 2015; Fernandez Turienzo, et al. 2020; Shen, et al. 2022; Swift, et al. 2021). In a meta-analysis study, education during pregnancy reported that women were prepared for pregnancy complications (Ketema, et al. 2020). Lack of information and fear of the unknown during pregnancy and birth increase the stress of pregnant women (Uludağ, et al. 2022).

These results emphasize the need for follow-up and education of pregnant women in order to reduce the negative effects on pregnant women after the earthquake. It is thought that individual training and pregnancy follow-up given to pregnant women in the earthquake zone in their living spaces will increase prenatal comfort and reduce the effects of distress, risk perception and birth anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak Turkish,
* First pregnancy
* Agreeing to participate in the study
* 14 weeks pregnant

Exclusion Criteria:

* Pregnant women who do not continue the program.
* Attending a pregnancy education class

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant
Enrollment: 64 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-12-09 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Prenatal Comfort Scale | hrough study completion, an average of 1 week
  The scale is evaluated out of a total of 75 points. It is interpreted that as the score decreases, the comfort level also decreases, and as the score increases, the comfort level also increases. The scale has no reverse-scored items and no cut-off points.
Prenatal Distress Scale | 15 minutes before the training, 15 minutes after the training is completed
  The total score of the items is taken as a value between 0-34. Yuksel et al. The cut-off value of the scale has not been calculated and a high score from the scale indicates a high level of prenatal distress.
Pregnancy Risk Perception Scale | 15 minutes before the training, 15 minutes after the training is completed
  Each item in the scale has a linear line of 0-10 cm (0-100 mm), and at the two ends of these lines are the expressions "no risk" and "extremely high risk". The total score of the scale is obtained by summing the scores of the nine items and dividing the resulting score by 9. A scoring can also be made for the factors of the scale: Similar to the total score calculation, it is calculated by dividing the sum of the scores from the relevant sub-dimensions of the scale by the number of items in that sub-dimension. The scale has no cut-off point. An increase in the score obtained from the scale indicates that the risk perception of the pregnant woman for herself and her baby increases.
Oxford Birth Anxiety Scale: | 15 minutes before the training, 15 minutes after the training is completed
  Women's concerns about the birth process were evaluated with a four-point Likert scale. Scale; It can be applied to women in all periods before, during and after birth; It was scored as "1: I was very worried", "2: I was quite worried", "3: I was not very worried", "4: I was not worried at all". The scale is evaluated based on the total score (min = 10, max = 40). It is interpreted that as the score increases, women's anxiety level decreases. The scale, which has three subscales: "pain and distress", "prenatal uncertainty" and "interventions", does not have reverse questions.

CONTACTS AND LOCATIONS:
Locations (1):
- TurkishMoHKahramanmarasPH, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Amarpoor Mesrkanlou H, Ghaemmaghami Hezaveh SJ, Tahmasebi S, Nikniaz Z, Nikniaz L. The Effect of an Earthquake Experienced During Pregnancy on Maternal Health and Birth Outcomes. Disaster Med Public Health Prep. 2022 Jun 27;17:e157. doi: 10.1017/dmp.2022.132. PMID 35757895
- [Background] Cankaya S, Simsek B. Effects of Antenatal Education on Fear of Birth, Depression, Anxiety, Childbirth Self-Efficacy, and Mode of Delivery in Primiparous Pregnant Women: A Prospective Randomized Controlled Study. Clin Nurs Res. 2021 Jul;30(6):818-829. doi: 10.1177/1054773820916984. Epub 2020 Apr 13. PMID 32281410
- [Background] Dennis CL, Dowswell T. Psychosocial and psychological interventions for preventing postpartum depression. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD001134. doi: 10.1002/14651858.CD001134.pub3. PMID 23450532
- [Background] Uludag E, Sercekus P, Vardar O, Ozkan S, Alatas SE. Effects of online antenatal education on worries about labour, fear of childbirth, preparedness for labour and fear of covid-19 during the covid-19 pandemic: A single-blind randomised controlled study. Midwifery. 2022 Dec;115:103484. doi: 10.1016/j.midw.2022.103484. Epub 2022 Sep 9. PMID 36155390
- [Background] Fernandez Turienzo C, Bick D, Briley AL, Bollard M, Coxon K, Cross P, Silverio SA, Singh C, Seed PT, Tribe RM, Shennan AH, Sandall J; POPPIE Pilot Collaborative Group. Midwifery continuity of care versus standard maternity care for women at increased risk of preterm birth: A hybrid implementation-effectiveness, randomised controlled pilot trial in the UK. PLoS Med. 2020 Oct 6;17(10):e1003350. doi: 10.1371/journal.pmed.1003350. eCollection 2020 Oct. PMID 33022010
- [Background] Gooijers J, Swinnen SP. Interactions between brain structure and behavior: the corpus callosum and bimanual coordination. Neurosci Biobehav Rev. 2014 Jun;43:1-19. doi: 10.1016/j.neubiorev.2014.03.008. Epub 2014 Mar 21. PMID 24661987
- [Background] Hawkins G, Gullam J, Belluscio L. The effect of a major earthquake experienced during the first trimester of pregnancy on the risk of preterm birth. Aust N Z J Obstet Gynaecol. 2019 Feb;59(1):82-88. doi: 10.1111/ajo.12797. Epub 2018 Mar 8. PMID 29516471
- [Background] Ketema DB, Leshargie CT, Kibret GD, Assemie MA, Petrucka P, Alebel A. Effects of maternal education on birth preparedness and complication readiness among Ethiopian pregnant women: a systematic review and meta-analysis. BMC Pregnancy Childbirth. 2020 Mar 6;20(1):149. doi: 10.1186/s12884-020-2812-7. PMID 32143581
- [Background] Kyozuka H, Murata T, Yasuda S, Ishii K, Fujimori K, Goto A, Yasumura S, Ota M, Hata K, Suzuki K, Nakai A, Ohira T, Ohto H, Kamiya K. The Effects of the Great East Japan Earthquake on Perinatal Outcomes: Results of the Pregnancy and Birth Survey in the Fukushima Health Management Survey. J Epidemiol. 2022;32(Suppl_XII):S57-S63. doi: 10.2188/jea.JE20210444. PMID 36464301
- [Background] Lian Q, Ni J, Zhang J, Little J, Luo S, Zhang L. Maternal exposure to Wenchuan earthquake and prolonged risk of offspring birth outcomes: a natural experiment study. BMC Pregnancy Childbirth. 2020 Sep 22;20(1):552. doi: 10.1186/s12884-020-03206-1. PMID 32962638
- [Background] Matvienko-Sikar K, Dockray S. Effects of a novel positive psychological intervention on prenatal stress and well-being: A pilot randomised controlled trial. Women Birth. 2017 Apr;30(2):e111-e118. doi: 10.1016/j.wombi.2016.10.003. Epub 2016 Oct 31. PMID 27810284
- [Background] Adal MN. The fine structure of the sensory region of cat muscle spindles. J Ultrastruct Res. 1969 Feb;26(3):332-53. doi: 10.1016/s0022-5320(69)80011-0. No abstract available. PMID 4237927
- [Background] O'Hara MW, Wisner KL. Perinatal mental illness: definition, description and aetiology. Best Pract Res Clin Obstet Gynaecol. 2014 Jan;28(1):3-12. doi: 10.1016/j.bpobgyn.2013.09.002. Epub 2013 Oct 7. PMID 24140480
- [Background] Palmeiro-Silva YK, Orellana P, Venegas P, Monteiro L, Varas-Godoy M, Norwitz E, Rice G, Osorio E, Illanes SE. Effects of earthquake on perinatal outcomes: A Chilean register-based study. PLoS One. 2018 Feb 23;13(2):e0191340. doi: 10.1371/journal.pone.0191340. eCollection 2018. PMID 29474413
- [Background] Silbereisen RK, Oesterreich R, Leitner K. [Configurations of attitudes, experiences and expectations of social welfare recipients]. Z Klin Psychol Psychother. 1977;25(3):256-63. German. PMID 595769
- [Background] Swift EM, Zoega H, Stoll K, Avery M, Gottfreethsdottir H. Enhanced Antenatal Care: Combining one-to-one and group Antenatal Care models to increase childbirth education and address childbirth fear. Women Birth. 2021 Jul;34(4):381-388. doi: 10.1016/j.wombi.2020.06.008. Epub 2020 Jul 24. PMID 32718800
- [Background] LeDoux JE, Wilson DH, Gazzaniga MS. A divided mind: observations on the conscious properties of the separated hemispheres. Ann Neurol. 1977 Nov;2(5):417-21. doi: 10.1002/ana.410020513. PMID 103484
- [Background] Watanabe Z, Iwama N, Nishigori H, Nishigori T, Mizuno S, Sakurai K, Ishikuro M, Obara T, Tatsuta N, Nishijima I, Fujiwara I, Nakai K, Arima T, Takeda T, Sugawara J, Kuriyama S, Metoki H, Yaegashi N; Japan Environment & Children's Study Group. Psychological distress during pregnancy in Miyagi after the Great East Japan Earthquake: The Japan Environment and Children's Study. J Affect Disord. 2016 Jan 15;190:341-348. doi: 10.1016/j.jad.2015.10.024. Epub 2015 Oct 28. PMID 26544618
- [Background] Yamashita K, Natsukawa T, Kubo T, Kondo H, Koido Y. Vulnerability of Pregnant Women After a Disaster: Experiences After the Kumamoto Earthquake in Japan. Prehosp Disaster Med. 2019 Oct;34(5):569-571. doi: 10.1017/S1049023X1900476X. Epub 2019 Aug 30. No abstract available. PMID 31466549
- [Background] Yuksel F, Akin S, Durna Z. Prenatal distress in Turkish pregnant women and factors associated with maternal prenatal distress. J Clin Nurs. 2014 Jan;23(1-2):54-64. doi: 10.1111/j.1365-2702.2012.04283.x. Epub 2013 Jan 11. PMID 23305376
- [Derived] Senol DK, Keles MG. The effect of individual education and care provided in living spaces to pregnant women in the earthquake region on prenatal distress, risk perception, and labour anxiety. BMC Pregnancy Childbirth. 2025 Feb 3;25(1):109. doi: 10.1186/s12884-025-07233-8. PMID 39901147